CLINICAL TRIAL: NCT02631395
Title: The Effect of a Shoulder Training Program to Prevent Shoulder Pain Among Girls in Junior Team Handball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SorTrondelagUC
Record Dates: First submitted 2015-05-05; First posted 2015-12-16 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Shoulder Pain
Keywords: Exercise movement techniques
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Other): Six teams, consisting of 13 to 25 players each, were randomized into two groups throughout their competition season; the training Group (intervention Group) and the Control Group.The intervention group completed strength training exercises Three times a week the Whole competition season.
  Interventions: Other: Exercise
- Control group (Other): The three teams in the Control Group trained as normal throughout the season and participated in a comparable handball training program, but did not conduct any specific upper--body strength training
  Interventions: Other: Control group

INTERVENTIONS:
Other: Exercise — Three teams participated in a seven--month, three--times--a--week shoulder--muscle strength--training program while three teams participated in a comparable handball training program but did not conduct any specific upper--body strength training.
  Arms: Training group
Other: Control group — The three teams in the Control Group trained as normal throughout the season and participated in a comparable handball training program, but did not conduct any specific upper--body strength training
  Arms: Control group

SUMMARY:
Very little is known about the potential for preventing the prevalence of shoulder complaints in handball players, particularly younger players. The aim of this study is to evaluate the effect of a shoulder training program on shoulder pain during a season of team handball.

DETAILED DESCRIPTION:
Six teams, consisting of 13 to 25 players each, were randomized into two groups throughout their competition seasons. Three teams participated in a seven--month, three--times--a--week shoulder--muscle strength--training program while three teams participated in a comparable handball training program but did not conduct any specific upper--body strength training. Effects of this strength--training program were evaluated by comparing pre-- and post--training data from a survey on shoulder complaints based on a self--report questionnaire (quick DASH) and Visual Analogue Scale (VAS). The players completed the VAS on pain once a month. In addition to that the players were tested in a maximum push up test, dynamometer test for internal and external rotation strength in the shoulder and throwing distance in the pre- and posttest.

ELIGIBILITY:
Inclusion Criteria:

- team handball players in the top division in the J16 class in the Trøndelag region in Norway

Exclusion Criteria:

- previous shoulder operations og fractures in the shoulder region

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Shoulder pain (Visual Analogue Scale) | 7 months
  Effects of this strength--training program were evaluated by comparing pre-- and post--training data from a survey on shoulder complaints based on a self--report questionnaire (quick DASH) and Visual Analogue Scale (VAS). The players completed the VAS form on shoulder pain in the beginning of the season, then once a month throughout the season, and then in the end of the season.

SECONDARY OUTCOMES:
Shoulder strength | 7 months
  External and internal rotation strength in the shoulder was measured with a handheld dynamometer in the beginning and in the end of the season.
Push ups | 7 months
  The Maximum number of push ups the players were able to perform was recorded in the beginning and in the end of the season.
Throwing distance | 7 months
  The Maximum throwing distance With a handball was recorded in the beginning and in the end of the season.
Shoulder function (Quick DASH) | 7 months
  The quick DASH questionaire was completed in the beginning and in the end of the season.
  In addition to the VAS and Quick DASH, the players were tested in a maximum push up test, dynamometer test for internal and external rotation strength in the shoulder and throwing distance in the pre- and posttest (see secondary outcome measures).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Harry Størksen, Study Director — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Osteras H, Sommervold M, Skjolberg A. Effects of a strength-training program for shoulder complaint prevention in female team handball athletes. A pilot study. J Sports Med Phys Fitness. 2015 Jul-Aug;55(7-8):761-7. Epub 2014 Dec 17. PMID 25514821